CLINICAL TRIAL: NCT03492658
Title: Abatacept to Silence Anti-citrullinated Protein Antibody-expressing B Cells in Rheumatoid Arthritis (ASCARA).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Hans Ulrich Scherer, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL62584.058.17
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis; Rheumatic Diseases
Keywords: abatacept; ACPA expressing B cells
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, single center, two-arm, investigator-initiated, interventional clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy (MTX/abatacept) (Experimental): Treatment with a combination of methotrexate (10 - 25 mg once weekly) and abatacept (125 mg subcutaneously once weekly) for 6 months, followed by methotrexate monotherapy (10 - 25 mg once weekly) for another 6 months.
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Methotrexate (MTX) monotherapy (Active Comparator): Treatment with methotrexate monotherapy (10 - 25 mg once weekly) for 12 months.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Abatacept — Patients will be randomized to treatment with either methotrexate monotherapy (10 - 25 mg once weekly) or a combination therapy of methotrexate (10 - 25 mg once weekly) and abatacept (125 mg subcutaneously once weekly) for 6 months, followed by methotrexate monotherapy (10 - 25 mg once weekly) in both groups for another 6 months.
  Other Names: Orencia
  Arms: Combination therapy (MTX/abatacept)
Drug: Methotrexate — Patients will be randomized to treatment with either methotrexate monotherapy (10 - 25 mg once weekly) or a combination therapy of methotrexate (10 - 25 mg once weekly) and abatacept (125 mg subcutaneously once weekly) for 6 months, followed by methotrexate monotherapy (10 - 25 mg once weekly) in both groups for another 6 months.

SUMMARY:
To investigate the effect of CTLA4-Ig (abatacept) on phenotype, transcriptional profile, B cell receptor usage and functional parameters of circulating B cells expressing anticitrullinated protein antibodies (ACPA) in patients with early, methotrexate-naïve, ACPA positive rheumatoid arthritis.

DETAILED DESCRIPTION:
B cells expressing anti citrullinated protein antibodies (ACPA) in patients with rheumatoid arthritis (RA) display an activated, proliferative phenotype. Experimental data indicate that ACPA and ACPA-expressing B cells are actively involved in driving the disease process in RA. The present study is based on the hypothesis that targeted intervention with CTLA4-Ig (abatacept) as a means to interfere with T cell help for B cells in early, active, ACPA-positive rheumatoid arthritis can reverse the activated, proliferative phenotype of citrullinated antigen-specific B cells.

ELIGIBILITY:
Inclusion Criteria:

Each patient must:

* have a diagnosis of rheumatoid arthritis according to the revised 2010 EULAR/ACR criteria for classification of RA
* have a positive test for the presence of anti-citrullinated protein antibodies (ACPA) in serum as determined by routine clinical assay.
* have adequate hematologic function (ANC ≥ 4000 cells/μL, platelet count ≥ 150000/μL, and hemoglobin ≥ 10 g/dL (corresponding to 6.2 mmol/L)
* have serum creatinine concentrations < 1.5 mg/dl and/or a normal creatinine clearance
* if a female patient is of childbearing potential, agree to: comply with effective contraceptive measures, use adequate contraception since the last menses, use adequate contraception during the study, have a negative pregnancy test within one week of study entry
* be willing to receive a booster vaccination against tetanus toxoid three to four weeks prior to randomization
* be able and willing to give written informed consent prior to entry in the study

Exclusion Criteria:

Any patient who has:

* been previously treated with either abatacept and/or methotrexate or another csDMARD
* been previously treated with a kinase inhibitor
* been previously treated with rituximab or another B-cell depleting agent
* been previously treated with a biological DMARD
* received intra-articular or systemic glucocorticoid injections or has required treatment for acute RA flare (not being part of a regular therapeutic regimen) within four weeks prior to randomization or requires narcotic analgesics other than those accepted by the investigator for analgesia (e.g. paracetamol, codeine, tramadol)
* been tested negative for anti citrullinated protein antibodies
* contraindications for a booster vaccination against tetanus toxoid prior to randomization to the treatment arms; if a patient refuses booster vaccination but has detectable numbers of tetanus toxoid-specific B cells circulating in peripheral blood prior to the baseline visit, the patient can still be allowed to participate in the study at the judgement of the investigator.
* evidence of any other major chronic inflammatory disease (i.e. psoriasis, psoriatic arthritis, spondyloarthritis or inflammatory bowel disease)
* evidence of poorly controlled diabetes, history of clinically significant pulmonary disease including interstitial lung disease or methotrexate-induced lung disease, poorly controlled asthma or a history of severe life-threatening asthma attacks, history of active tuberculosis, history of latent tuberculosis without adequate medical treatment, liver cirrhosis or fibrosis, significant active infection or any underlying diseases that could predispose the subject to infections
* liver function abnormality (total bilirubin ≥ 1.5x the upper limit of normal range, AST, ALT ≥ 3x upper limit of normal range)
* concurrent treatment with an experimental drug or who has participated in another clinical trial with an investigational drug within 30 days prior to study entry
* pre-existing sensory or motor polyneuropathy ≥ Grade 2 according to NCI CTC
* past or current history of neoplasms, except for curatively treated non-melanoma skin cancer, adequately treated in situ carcinoma of the cervix or another cancer curatively treated and with no evidence of disease for at least 10 years
* significant cardiac disease, cardiac arrhythmia (Lown Grade ≥ III), uncontrolled hypertension or recent history of myocardial ischemia
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Percentage of ACPA-expressing B cells that express the marker Ki-67 | 24 weeks
  Flow cytometry-based determination of the percentage of ACPA-expressing B cells that stain positive for Ki-67, circulating in peripheral blood of patients with early, ACPA-positive rheumatoid arthritis.

SECONDARY OUTCOMES:
Change in disease activity | 24 weeks
  The change from baseline in disease activity (expressed as DAS 44).

OTHER OUTCOMES:
Percentage of patients achieving remission | 12, 24, 36 and 48 weeks
  To evaluate the percentage of patients achieving SDAI remission.
Monitor treatment-related immunological serum/plasma markers | Each study visit: baseline + 12, 24, 36 and 48 weeks
  to monitor treatment-related immunological serum/plasma markers (rheumatoid factor (IgM), anti-citrullinated protein antibodies and antibodies against other posttranslational modified proteins (AMPAs), anti-tetanus toxoid antibodies, IgG, IgA, IgM, and phenotypic cellular markers on circulating lymphocytes.
Change of expression level the marker Ki-67 | 12, 36 and 48 weeks
  Evaluate the change of expression level (from baseline) of the marker Ki-67 on memory B cells expressing ACPA versus memory B cells specific for recall antigens (tetanus toxoid) in peripheral blood.
Change in serum/plasma parameters related to disease activity | 12, 24, 36 and 48 weeks
  Evaluate the change from baseline in serum/plasma parameters related to disease activity (e.g. erythrocyte sedimentation rate, C-reactive protein, interleukin-6, -8, -10, TNF-alpha, vascular endothelial growth factor, granulocyte-monocyte colony stimulating factor).
Change of expression level of the markers CD80, CD86 and HLA-DR | 12, 24, 36 and 48 weeks
  Evaluate the change of expression level (from baseline) of the markers CD80, CD86 and HLA-DR on memory B cells expressing ACPA versus memory B cells specific for recall antigens (tetanus toxoid) in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Ulrich Scherer, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Willemze A, Trouw LA, Toes RE, Huizinga TW. The influence of ACPA status and characteristics on the course of RA. Nat Rev Rheumatol. 2012 Jan 31;8(3):144-52. doi: 10.1038/nrrheum.2011.204. PMID 22293763
- [Background] Keating GM. Abatacept: a review of its use in the management of rheumatoid arthritis. Drugs. 2013 Jul;73(10):1095-119. doi: 10.1007/s40265-013-0080-9. PMID 23794171
- [Background] Kerkman PF, Fabre E, van der Voort EI, Zaldumbide A, Rombouts Y, Rispens T, Wolbink G, Hoeben RC, Spits H, Baeten DL, Huizinga TW, Toes RE, Scherer HU. Identification and characterisation of citrullinated antigen-specific B cells in peripheral blood of patients with rheumatoid arthritis. Ann Rheum Dis. 2016 Jun;75(6):1170-6. doi: 10.1136/annrheumdis-2014-207182. Epub 2015 Jun 1. PMID 26034045